CLINICAL TRIAL: NCT00006112
Title: Randomized Therapeutic Study Comparing Tumor Resection Followed Immediately by Intraperitoneal Chemotherapy and Systemic Chemotherapy VS Systemic Chemotherapy Alone for the Treatment of Colorectal Cancer Metastatic to the Peritoneum
Brief Title: Fluorouracil With or Without Mitomycin in Treating Patients With Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068124; FRE-IGR-95/040/434-SUGAR; EU-20012
Record Dates: First submitted 2000-08-03; First posted 2004-05-04 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2001-05

CONDITIONS: Carcinoma of the Appendix; Colorectal Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; carcinoma of the appendix; primary peritoneal cavity cancer
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Drug Therapy; Fluorouracil; Leucovorin; Mitomycin

INTERVENTIONS:
Drug: chemotherapy
Drug: fluorouracil
Drug: leucovorin calcium
Drug: mitomycin C

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of fluorouracil with or without mitomycin in treating patients who have peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of adjuvant systemic fluorouracil with intraperitoneal mitomycin vs systemic fluorouracil alone in terms of survival in patients with peritoneal cancer originating from the colorectum.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center and mode of surgery. Patients are randomized to one of two treatment arms. Arm I: Patients undergo complete resection of tumor on day 0. Patients then receive mitomycin intraperitoneally (IP) over 23 hours on day 1 and fluorouracil IP over 24 hours on days 2-5. Patients then receive one of three systemic chemotherapy regimens for 6 months: Regimen I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 22 hours on days 1 and 2. Treatment repeats every 2 weeks. Regimen II: Patients receive fluorouracil IV continuously for 7 weeks. Treatment repeats every 8 weeks. Regimen III: Leucovorin calcium and fluorouracil are administered as per standard procedure. Arm II: Patients receive treatment as in arm I but without early intraperitoneal chemotherapy. Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: At least 90 patients (45 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven peritoneal cancer that is amenable to total resection Originated as colorectal adenocarcinoma or cancer of the appendix No diffuse (unresectable) tumors No microscopic cancer only No hepatic, lymph node, or extraabdominal metastases on the preoperative work-up No primitive peritoneal mesothelioma No peritoneal pseudomyxomas or ascites No cancer that originates as ovarian or neuroendocrine cancer, especially sarcomas (intra- or retroperitoneal) Complete resection of tumor deposit No originating cancer of unknown origin

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC greater than 1,500/mm3 Platelet count greater than 100,000/mm3 No chronic hematologic disorder No coagulation disorder Hepatic: Not specified Renal: Creatinine less than 1.36 mg/dL Other: No significant medical condition that would preclude study

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Elias, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France